CLINICAL TRIAL: NCT00846495
Title: A Randomized, Single-Blind Pilot Study to Compare the Efficacy and Cost-Effectiveness of Frovatriptan vs. Topiramate for the Prevention of Migraine
Brief Title: Pilot Study to Compare Frovatriptan vs. Topiramate for Prevention of Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinvest (Individual)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Clinvest, CEO, Cady, Roger, M.D.
Organization: Cady, Roger, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Frova vs. Topiramate
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Migraine
Keywords: Migraine; Migraine prevention; Prodrome; Premonitory phase; Preemptive therapy
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate; frovatriptan

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- topiramate (Active Comparator): Subjects randomized to Group A at Visit 2 were provided with topiramate, titrated over 4 weeks to a maximum dose of 100 mg daily. One dosage adjustment was allowed with a minimum dose of 50 mg daily.
  Interventions: Drug: topiramate
- frovatriptan (Active Comparator): Subjects randomized to Group B at Visit 2 were provided with frovatriptan 5 mg to treat during prodrome at the point they were confident a disabling migraine would occur (before the onset of headache).
  Interventions: Drug: frovatriptan

INTERVENTIONS:
Drug: topiramate — topiramate 25mg 1 tab in PM x 1 week topiramate 25mg 1 tab in AM / 1 tab in PM x 1 week topiramate 25mg 1 tab in AM / 2 tabs in PM x 1 week topiramate 25mg 2 tabs in AM / 2 tabs in PM x 5 weeks
  Other Names: Topamax
  Arms: topiramate
Drug: frovatriptan — frovatriptan 5mg tab during premonitory phase of migraine
  Other Names: Frova
  Arms: frovatriptan

SUMMARY:
Subjects enrolled at 2 investigative sites will complete 3 visits. Following Visit 1, during a 1-month Baseline Period, subjects will treat with their usual medication and document any warning signs (Prodrome pre-headache) that a migraine will occur. Following randomization (like a flip of the coin) at Visit 2, subjects will treat daily with topiramate or during Prodrome with frovatriptan. Subjects complete a 2-month Treatment Period before exit at Visit 3.This study will compare the effectiveness of daily treatment vs. treatment during the pre-headache phase for prevention of migraine.

ELIGIBILITY:
INCLUSION CRITERIA

1. Subject has at least a one-year history of migraine with or without aura meeting International Headache Society criteria (see Appendix)
2. Subject has a 3-month history of averaging 3-6 migraines per month
3. Subject reports premonitory symptoms and the ability to predict at least 50% of high impact headaches
4. Subjects must currently or have in the past successfully utilized a triptan as an acute treatment for migraine as determined by the investigator.
5. Male or female at least 18 years of age
6. Subject of childbearing potential agrees to use adequate contraception during the study. Adequate methods of contraception are to be determined by the investigator and should be consistent with contraceptive care administered in the regular clinical use of frovatriptan and topiramate.
7. Subject is aware of prodrome symptoms that may include physiological, psychological or cognitive changes. These may include, but are not limited to such symptoms as Pre-Menstrual Syndrome (PMS), change in mood, energy level, appetite, food craving, nausea, sense of hearing, sense of smell or swelling/fluid retention, excessive yawning, head pain, muscle pain/tenderness, irritability, confusion, extreme sleepiness, impaired speech or impaired memory. (The subject should be able to differentiate these symptoms from other similar symptoms that do not precede migraine). The symptoms should precede migraine by 4-24 hours signaling an impending migraine attack.
8. Subject is able to understand instructions for the study and complete the diary
9. Subject is willing to give informed consent to participate in the study
10. Any migraine prophylactic medication must have a stabilized dosage for one month

EXCLUSION CRITERIA

1. History of any medical condition that would confound the results of the study including but not limited to the following:

   * Hepatic disease or significant hepatic dysfunction
   * History of pancreatitis
   * History of thrombocytopenia
   * History of glaucoma
   * History of osteoporosis or osteopenia
   * Cardiovascular Disease - Coronary artery disease, Ischemic heart disease or Significant Arrhythmia
   * History of active Cerebrovascular Disease
   * Hypertension - Uncontrolled hypertension in a non-migrainous state (> 160 mmHg systolic or >95 mmHg. diastolic). Hypertension must be controlled effectively with medication for a period of 3 months.
   * Basilar or Hemiplegic Migraine
   * Significant peripheral vascular disease or Raynaud's Syndrome
   * Significant Active Renal, Hepatic, Gastrointestinal, Endocrine or
   * Neurological Disease
   * History of depression, mood problems or suicidal thoughts or behavior that in the opinion of the Investigator would interfere with participation in the study.
2. History of ergotamine, "triptan", or analgesic abuse within past 3 months
3. History of current or recent drug or alcohol abuse that would interfere with participation in the study.
4. More than 15 headache days per month within past 3 months.
5. Women who are pregnant or breast feeding
6. Subjects with known hypersensitivity or intolerance to topiramate or any triptan-like medication
7. Subject is scheduled for surgical procedure to occur while enrolled in study.that in opinion of the Investigator would interfere with participation in the study.
8. Subject is on a ketogenic diet
9. Participation in another investigative drug study within the previous 30 days
10. Excluded medications: MAO Inhibitors, lithium, methylergonovine, methysergide, ergotamine-containing products, or topiramate daily for migraine prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Principal Investigator — Clinvest
Locations (2):
- United States (2):
  - Physician Associates LLC, Oviedo, Florida
  - Clinvest, Springfield, Missouri

REFERENCES:
- [Background] Luciani R, Carter D, Mannix L, Hemphill M, Diamond M, Cady R. Prevention of migraine during prodrome with naratriptan. Cephalalgia. 2000 Mar;20(2):122-6. doi: 10.1046/j.1468-2982.2000.00030.x. PMID 10961768

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate: Subjects randomized to Group A were provided with topiramate 25mg to titrate to a maximum dosage of 100mg during Month 1. One dose adjustment was allowed with 50mg/day the required minimum dosage. Group A subjects treated with daily topiramate during Months 2 and 3 and rescued any migraine headache that occurred with frovatriptan 2.5mg.
- Frovatriptan: Subjects randomized to Group B were provided with frovatriptan 5mg to be utilized during prodrome at the point they were confident a disabling migraine would occur but before the onset of headache. Subjects were provided with frovatriptan 2.5mg for rescue of persistent or recurring headache between 4 and 24 hours following treatment during prodrome.
Period: Overall Study
Arm/Group | Topiramate | Frovatriptan
Started | 28 | 27
Completed | 20 | 24
Not Completed | 8 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 5 | 1
Not completed — Lack of Efficacy | 1 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Frovatriptan | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 27 | 55
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.61 (10.3) | 37.33 (9.46) | 37.47 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Migraine Attacks in Participants Using Frovatriptan in a Preemptive Treatment Paradigm vs. Daily Topiramate
Description: Compare number of migraine attacks reported by participants using frovatriptan in a preemptive treatment paradigm vs. daily topiramate during Treatment Period Month 2
Time Frame: Treatment Month 2
Population: Number of Units Analyzed is equivalent to number of migraine attacks reported during 2nd Treatment Month.
Measure: Mean (Standard Deviation); unit: Migraine attacks
Units Other Than Participants: Migraine attacks
Arm/Group | Topiramate | Frovatriptan
Number analyzed (Participants) | 20 | 24
Number analyzed (Migraine attacks) | 27 | 51
Migraine attacks | 1.35 (1.31) | 2.12 (1.75)

2. Primary Outcome: Number of Headache Days Reported by Participants Using Frovatriptan in a Preemptive Treatment Paradigm vs. Daily Topiramate to Prevent Migraine
Description: Measure the change in number of headache days between participants using frovatriptan in a preemptive treatment paradigm vs. daily topiramate to prevent migraine
Time Frame: Treatment Month 2
Measure: Mean (Standard Deviation); unit: Headache Days
Arm/Group | Topiramate | Frovatriptan
Number analyzed (Participants) | 20 | 24
Headache Days | 4.75 (2.59) | 2.79 (3.26)

3. Secondary Outcome: Number of Headache Days Each Month Following Initiation of Treatment With Study Medication
Description: Measure the change in number of headache days reported by participants during each treatment month following initiation of treatment with study medication
Time Frame: 2 Months
Population: Number of Units Analyzed is equivalent to number of headache days reported during Treatment Months 1 and 2.
Measure: Mean (Standard Deviation); unit: Headache Days
Units Other Than Participants: Headache Days
Arm/Group | Topiramate | Frovatriptan
Number analyzed (Participants) | 20 | 24
Number analyzed (Headache Days) | 119 | 177
Headache Days
  Treatment Month 1 | 4.20 (2.88) | 3.96 (2.84)
  Treatment Month 2 | 1.75 (1.86) | 3.42 (2.98)

4. Secondary Outcome: Participants With Greater Than 50% Reduction in Migraine Attacks and Headache Days Per Month Utilizing Each Treatment Paradigm
Description: Compare number of participants with greater than 50% reduction in migraine attacks and headache days from Baseline to Treatment Months 1 and 2
Time Frame: 2 Months
Measure: Number; unit: Participants
Arm/Group | Topiramate | Frovatriptan
Number analyzed (Participants) | 20 | 24
Participants
  Migraine Attacks Treatment Month 1 | 11 | 13
  Headache Days Treatment Month 1 | 7 | 9
  Migraine Attacks Treatment Month 2 | 15 | 15
  Headache Days Treatment Month 2 | 16 | 13

5. Secondary Outcome: Quality of Life in Subjects Utilizing Each Treatment Paradigm
Description: Quality of Life is measured by the Migraine Specific Quality of Life Questionnaire (MSQ), which includes 3 dimensions: Role Function Restrictive (degree to which performance of daily activities is limited), Role Function Preventive (degree to which performance of daily activities is interrupted), and Emotional Function (frustration and helplessness due to migraine). Scores range from 0 to 100. For each dimension, a higher score indicates a better health status. Participants completed the MSQ at Randomization, and after Treatment Months 1 and 2.
Time Frame: Randomization, End of Treatment Month 1, End of Treatment Month 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Topiramate | Frovatriptan
Number analyzed (Participants) | 20 | 24
Score on a Scale
  Role Function Restrictive - Baseline | 56.00 (15.88) | 59.88 (16.65)
  Role Function Restrictive - Treatment Month 1 | 80.29 (19.33) | 66.48 (18.75)
  Role Function Restrictive - Treatment Month 2 | 86.64 (13.98) | 71.84 (19.57)
  Role Function Preventive - Baseline | 77.75 (16.02) | 77.50 (18.53)
  Role Function Preventive - Treatment Month 1 | 85.25 (18.32) | 79.25 (21.96)
  Role Function Preventive - Treatment Month 2 | 93.95 (7.57) | 84.96 (16.67)
  Emotional Function - Baseline | 60.67 (22.47) | 64.71 (23.13)
  Emotional Function - Treatment Month 1 | 80.00 (25.68) | 73.18 (21.59)
  Emotional Function - Treatment Month 2 | 91.46 (10.49) | 75.10 (24.04)

6. Secondary Outcome: Participant Satisfaction With Study Medications
Description: Participant satisfaction is measured by the Patient Perception of Migraine Questionnaire (PPMQ). Questions were categorized within 6 dimensions: Efficacy, Functionality, Ease of Use, Cost, Bothersomeness of Side Effects, and Total Score. Scores range from 0 to 100. Higher scores represent better satisfaction.
  Participants completed the PPMQ 24 hours following each first dose of frovatriptan.
Time Frame: Treatment Month 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Topiramate | Frovatriptan
Number analyzed (Participants) | 20 | 24
Score on a Scale
  Efficacy | 76.7857 (21.04) | 75.1977 (30.21)
  Functionality | 77.8214 (22.68) | 76.3648 (29.98)
  Ease of Use | 91.6607 (11.5639) | 92.6989 (11.36)
  Cost | 81.2536 (19.85) | 59.0886 (32.86)
  Bothersomeness of Side Effects | 95.1786 (6.08) | 95.5398 (6.81)
  Total Score | 82.0925 (15.77) | 81.1417 (21.76)

7. Secondary Outcome: Adverse Events Associated With Study Medications
Description: Includes Adverse Events at or above 5% frequency per group.
Time Frame: Treatment Months 1 and 2
Measure: Number; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Topiramate | Frovatriptan
Number analyzed (Participants) | 20 | 24
Number analyzed (Adverse Events) | 45 | 43
Adverse Events | 26 | 11

8. Secondary Outcome: Cost of Frovatriptan vs. Topiramate as Preventive Treatment of Migraine
Description: Average cost of study medication taken by each subject. Measured in dollars.
Time Frame: Treatment Months 1 and 2
Measure: Mean (Standard Deviation); unit: Dollars (US)
Arm/Group | Topiramate | Frovatriptan
Number analyzed (Participants) | 20 | 24
Dollars (US)
  Preventive Medication Taken | 343.56 (50.4774) | 101.41 (10.304)
  Rescue Medication Taken | 38.33 (10.45) | 59.94 (9.54)
  All Study Medication Taken | 381.89 (51.8816) | 161.35 (70.1844)

ADVERSE EVENTS:
Arm/Group | Topiramate | Frovatriptan
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 17/28 | 5/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=28) | Frovatriptan (N=27)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Cold Symptoms (General disorders) | 0 (0) | 2 (2)
Concentration Problems (General disorders) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Dizziness (General disorders) | 1 (1) | 2 (3)
Irritability (General disorders) | 2 (2) | 0 (0)
Memory Problems (General disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Numbness in Extremities (Nervous system disorders) | 2 (2) | 0 (0)
Stomach Flu (Gastrointestinal disorders) | 2 (2) | 0 (0)
Taste Aversion (General disorders) | 3 (3) | 0 (0)
Tingling in Extremities (Nervous system disorders) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No